# 知情同意书

经皮穴位电刺激对全身麻醉下行腹部手术的老年患者术后 谵妄及脑电图特征参数的影响:单中心、随机、双盲、平行 对照临床试验

研究中心: 西京医院

主要研究者: 路志红

版本号: V1.0

版本日期: 2022年09月20日

# 知情同意书告知页

亲爱的患者:

诚邀您参加一项经皮穴位电刺激对全身麻醉下行腹部手术的老年患者术后 谵妄及脑电图特征参数的影响的临床试验性研究。在您同意参加该项试验之前, 请您仔细阅读这份知情同意书,它可以帮助您了解该项研究以及为何要进行这项 研究,研究的程序和期限,参加研究后可能给您带来的益处、风险和不适。如果 您愿意,您也可以和您的亲属、朋友一起讨论,帮助您做出决定,并向您的研究 人员提出任何您需要了解的问题,直至得到满意的答复。如果您同意参加本研究, 请您签署此知情同意书,并保存该份经您和研究者双方签字的知情同意书的复印 件。

## 研究目的和背景

本研究的目的是探究 TEAS 对全身麻醉下行腹部手术老年患者术后谵妄及其机制的影响,以验证 TEAS 能否改善腹部手术老年患者 POD 的发生率。

本研究将在西京医院麻醉科进行,预计至少有 226 名受试者自愿参加,本中 心预计完成 226 例。

空军军医大学第一附属医院(西京医院)伦理委员会已经审查并批准此项研究,认为此项研究符合是我国相关法律、法规要求,遵从赫尔辛基宣言原则,符合涉及人类的生物医学研究伦理指导原则的。

在全球性人口老龄化的背景下,当前我国人口老龄化已成为人口发展的常态,并且人口老龄化的速度明显加快,程度持续加深。随着人口老龄化发展,接受全身麻醉手术治疗的老年患者比例不断增加,老年患者(即 65 岁或以上)是合并术后谵妄(postaction delirium, POD)的高危人群,POD 是一种以注意力不集中、思维紊乱和意识水平改变为特征的一过性脑功能障碍综合征,通常发生于术后数小时至数日内。高龄是 POD 的独立危险因素,根据不同的研究人群和手术类型,POD 发生率为 20%~80%。POD 不仅会造成住院时间延长,术后并发症增加,甚至会造成永久性的认知功能损害,降低患者的远期生存率和生活质量。由于谵妄发生的机制尚不清楚,缺乏有效的治疗策略,因此,预防谵妄的发生发展至关重要。

脑电图(electroencephalogram, EEG)及脑电相关指标是反映大脑意识状态的重要指标,不同麻醉药物及麻醉深度引起不同的 EEG 特征性变化。研究表明,原始 EEG 与 POD 的发生发展有一定的相关性,并具有潜在的预测 POD 的价值。例如,心脏手术全麻期间较低的前额叶α波段功率与较差的术后认知功能有关,患者年龄越大 EEG 的特征性改变与 POD 的发生越显著。一项在老年人腹部手术中进行的研究也进一步证实了术中 EEG 低α功率与 POD 有关。此外,最近的一项研究表明,闭眼状态时枕部的α波段相对功率具有中等的辨别能力,与谵妄严重程度和注意力不集中严重程度成反比。

经皮穴位电刺激( transcutaneous electrical acupoint stimulation, TEAS)疗法是一种新型物理治疗方法,其将电神经疗法与中医针灸穴位相结合,通过穴位将低频脉冲电流输入,在进行穴位刺激的同时施行低频电疗,以达到治疗疾病的目的。中医认为手少阴心经与手厥阴心包经主情志,用于增强睡眠,治疗神经类疾病。神门穴是手少阴心经的穴位之一,有帮助入眠,调节自律神经,补益心气,安定心神等功效;内关穴是手厥阴心包经的常用腧穴之一,可调节神志,治疗神经衰弱、失眠、中风及后遗症。既往研究显示, TEAS 刺激双侧内关、神门穴可改善老年髋部手术患者围术期睡眠质量和减少术后谵妄发生率,而对于老年腹部手术患者的研究证据是十分有限的,TEAS 改善 POD 的机制也尚未明确,其伴随的脑电生物标志物及脑电深度变化仍需进一步的探索。因此,应特别加强对老年腹部手术患者围术期脑电活动的监测,以期通过对 EEG 的分析给 TEAS 对 POD 改善提供一个强有力的证据。

故本研究旨在观察 TEAS 内关、神门穴改善围术期老年患者 POD 并伴随某些特定脑电参数的变化,从而进一步探究 TEAS 的作用机制。

#### 哪些人不宜参加此项研究

#### 入选标准为:

- (1) 年龄>65 周岁;
- (2) 拟行全身麻醉下择期腹部手术患者;
- (3) ASA≤Ⅲ级;
- (4) 手术时长>2h:

- (5) 住院时长>3d;
- (6) 签署知情同意书。

#### 排除标准为:

- (1) 有严重中枢神经系统损伤及严重脑血管疾病患者(格拉斯哥-匹兹堡脑功能表现分级(cerebral performance category, CPC)评分 3~5 级);
- (2) 术前谵妄评定(CAM)阳性;
- (3) 无法配合研究者,如精神疾病或语言障碍;
- (4) 严重的肝肾功能不全 (Child-Pugh 肝功能分级 B、C 级、血肌酐>186 μ mol/L):
- (5) 呼吸衰竭(包括 I 型呼衰和 II 型呼衰)、COPD、支气管扩张症、肺结核等严重的呼吸系统疾病;
- (6) 不适宜实施经皮穴位电刺激者,如体内植入电生理装置、穴位部位皮肤 感染破损者。

## 研究设计和步骤

本研究为前瞻性随机对照临床研究。如果您符合入选条件并愿意参加该项研究的话,您将会被随机分到经皮穴位电刺激组和对照组。经皮穴位电刺激组将接经皮穴位电刺激干预;对照组将不接受任何干预。对两组均进行脑电图及脑氧饱和度监测,其余麻醉用药和监测均按临床常规方法实施。

#### 可能的风险与不适

本研究所采用干预措施为经皮穴位电刺激,为临床常用的穴位电刺激法,可能的风险均为常规麻醉和手术的风险。

如果在研究中您出现任何不适,请及时通知研究者,他/她将对此作出判断和医疗处理。

## 受试者保护及相关费用

在整个试验研究过程中,我们将严格遵守保护受试者的原则,将维护受试者的安全置于首要地位。

本研究对您无经济补助。所用麻醉方案为临床常用麻醉方案,费用由受试者 自行承担。如果从进入本项研究开始到试验持续的时间内,您发生了由学术委员 会和伦理委员会判定与本研究有关的损失,将获得相应补偿;若您发生了由学术委员会和伦理委员会判定与本研究有关的损伤,您将及时获得治疗,并按照中国的法律法规对您进行相应的赔偿。

## 可能的受益

您和其他受试者参与本研究所得到的临床结果,有可能会对老年手术中麻醉管理的优化做出贡献。

## 您的权益

您参加本研究是完全自愿的,因此您可以在任何时候决定退出研究。您不会 因此受到歧视或遭受利益损失。您的退出不会影响您和研究者的关系。并且您做 出的这一决定不会给您带来不利的影响,也不会妨碍您接受其他治疗。

如果您对本研究有任何问题,包括对受试者权益或对治疗处理措施方面的疑问,您可以随时直接与负责本研究的医生联系(路志红,029-84775343)。您有权随时了解与您有关的信息资料,研究人员将尽量详细回答您的每个问题和与研究相关事宜的咨询。

## 保密

您的研究记录(研究病历、检查报告等)将完整地保存在西京医院麻醉科。 您的信息在任何时候都会被保密。只有研究医生保留您的基本信息,在研究的其 他文件中将使用您的姓名缩写和代码标识。除了您的研究医生外,本研究的申办 科室代表,监察员、伦理委员会的代表可能将会查阅您与本研究有关的原始医疗 资料以确保研究是规范的,数据是真实可靠的。但所有的信息将会保密,本研究 结果可能会发表在医学杂志上,但也不会泄露您的身份。任何有关本项研究结果 的公开报告将不会披露您的个人身份。我们将在法律允许的范围内,尽一切努力 保护您个人医疗资料的隐私。

除本研究以外,有可能在今后的其他研究中会再次利用您的研究记录。您现在也可以声明拒绝除本研究外的其他研究利用您的医疗记录和病理标本。

#### 怎样获得更多的信息?

您可以在任何时间提出有关本项研究的任何问题。您的研究者将给您留下他/她的电话号码以便能回答您的问题。如果在研究过程中有任何重要的新信息,可能影响您继续参加研究的意愿时,您的研究者将会及时通知您。

#### 自主参加原则

您参加本研究完全是自愿的。您有权随时退出研究而不会遭到歧视或报复,您的权益也不会受到影响。您有权了解有关研究可能带来的不良反应。若继续参加本研究会对您的健康造成损害,或您的健康已不适合继续参加试验,或您不能遵守实验方案的要求,您的研究医生可以终止您的研究而不必得到您的同意。如果您决定退出研究,请您务必与路志红医生联系,将会对您进行各项指标的评估。

#### 现在该做什么?

是否参加本项研究由您自己决定。您可以和您的家人或朋友讨论后再做出决定。在您做出参加研究的决定前,请尽可能向研究者询问有关问题,直至您对本项研究完全理解。

该试验方案经医院伦理委员会批准实施,试验过程中有任何违反研究方案的情况,您可以直接向医院伦理委员会投诉。联系电话:029-84771794,电邮:xjyyllwyh@163.com。

## 受试者知情同意签字页

我已详细阅读了以上知情同意书,并理解了研究的目的以及参加研究的可能 受益和风险。研究者已将以上医学术语作了明确解释。我有机会提出问题并且所 有问题均得到了通俗易懂的答复。我可以选择不参加本项研究,或在任何时候通 知负责医生后退出,我的任何医疗待遇与权益不会因此而受到影响。如果我需要 其他治疗,或者我没有遵守研究计划,或者发生了与研究相关的损伤,或者有任 何其他原因,负责医生可以终止我继续参与本项研究。

我已阅读了以上知情同意书并获得副本,我的医师也向我作了详尽的说明。 我自愿参加本次临床试验。我同意有关方面对照我的原始医疗记录,检查核对试验研究收集的资料。

| 受试者正楷姓名: | 受试者电话: | |
|----------------------------------|--------------|-------------|
| 受试者签名: | 日期: | (年/月/日/) |
| (注:受试者无民事行为能力时<br>受试者及其监护人需要签名) | ,需监护人签名;受试者为 | 为限制民事行为能力时, |
| 监护人正楷姓名: | 与受试者关系: | |
| 监护人签名: | 监护人电话: | |
| 日期:(年 | 4月/日) | |
| 我确认已向病人详尽解释了》<br>风险,并解答了患者提出的所有[ | | 括病人可能的获益和 |
| 研究者签名(正楷): | 日期: | (年/月/日) |
| 研究者由话: | 日期. | (年/日/日) |